CLINICAL TRIAL: NCT05487677
Title: Augmentation of Subscapularis Repair in Total Shoulder Arthroplasty
Brief Title: Subscapularis Repair Augmentation for Total Shoulder Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael T. Freehill, Associate Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64618
Record Dates: First submitted 2022-07-22; First posted 2022-08-04 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: Patients undergoing reverse shoulder arthroplasty will be recruited, consented, & enrolled. Patient will be randomized to standard repair with sutures versus standard repair with BioBrace augmentation of the repair.
Who Masked: Participant, Outcomes Assessor
Masking Description: The physician performing the ultrasound evaluation will be blinded to which treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BioBrace Augmentation (Experimental): During the shoulder replacement surgery (arthroplasty) in order to access the shoulder, the subscapularis is removed from its insertion in your upper arm bone. It is repaired in reverse total shoulder arthroplasty, but is sometimes not as robust as we would like based on tissue quality and other factors. A shoulder arthroplasty is when the ball and socket are replaced with prosthetic components. If randomized to the BioBrace, patient will receive BioBrace augmentation of the standard subscapularis repair.
  Interventions: Device: BioBrace Augmentation
- Standard Repair with Sutures (Active Comparator): During the shoulder replacement surgery (arthroplasty) in order to access the shoulder, the subscapularis is removed from its insertion in your upper arm bone. It is repaired in reverse total shoulder arthroplasty, but is sometimes not as robust as we would like based on tissue quality and other factors. A shoulder arthroplasty is when the ball and socket are replaced with prosthetic components. If randomized to standard repair, patient will receive the standard repair with sutures.
  Interventions: Procedure: Standard Repair with Sutures

INTERVENTIONS:
Device: BioBrace Augmentation — During shoulder replacement surgery, the subscapularis (rotator cuff muscle) is sometimes repaired back again. This will be stitched and augmented with a BioBrace. The Biobrace is a biocomposite scaffold meaning both synthetic and biologic, compared to other traditional implants that are either synthetic or biologic. The stitch in the BioBrace group will be anchored to and reinforced by this material.
  Other Names: Implant Group
  Arms: BioBrace Augmentation
Procedure: Standard Repair with Sutures — During shoulder replacement surgery, the Subscapularis (rotator cuff muscle) is sometimes repaired back again. This is usually repaired with stitches per standard of care treatment.
  Other Names: Stitch Group
  Arms: Standard Repair with Sutures

SUMMARY:
The primary purpose of this research is to compare the images obtained by ultrasound between a standard repair of the subscapularis tissue and after repair with a Biobrace. The secondary purpose is to determine if there are any clinical differences.

DETAILED DESCRIPTION:
The investigators would like to learn if subscapularis repair augmentation with the Biobrace in total shoulder arthroplasty (reverse and anatomic) will result in sonographic and/or clinical improvements. This will allow for improvements in technique and better outcomes for patients going forward.

ELIGIBILITY:
Inclusion Criteria:

* Total Shoulder Arthroplasty

Exclusion Criteria:

* Vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in continuity of subscapularis tissue on ultrasound | 6 weeks, 6 months after surgery
  Continuity of subscapularis tissue on ultrasound
Difference in thickness of the subscapularis tissue on ultrasound | 3 months, 1 years after surgery
  Thickness of subscapularis tissue on ultrasound
Evaluate arthritis on shoulder x-ray | Surgery
  Amount of arthritis or wear patterns on shoulder x-Ray
Difference in signs of loosening or wear patterns in shoulder X-Ray | 2 weeks, 3 months, 6 months, 1 year, 2 years after surgery
  Signs of loosening or wear patterns on shoulder x-ray

SECONDARY OUTCOMES:
American Shoulder & Elbow Surgeons Score (ASES) score | 2 weeks, 3 months, 6 months, 1 year, 2 years after surgery
  is a 100-point scale that consists of two dimensions: pain and activities of daily living. 0 indicates worse shoulder condition and 100 indicates best shoulder condition. The greater the score, the lower the level of shoulder disability
Shoulder examination for the difference in Passive Range of Motion | 2 weeks, 3 months, 6 months, 1 year, 2 years after surgery
  Examining passive range of motion - forward flexion, external rotation, abduction
Shoulder examination for the difference in Active Range of Motion | 3 months, 6 months, 1 year, 2 years after surgery
  Examining active range of motion - internal rotation up posterior thorax. Strength- Jobes, external rotation, lift-off and belly-press

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Freehill, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States